CLINICAL TRIAL: NCT06668337
Title: A Randomized Controlled Trial Comparing the Effectiveness of Different Doses of Ephedrine Infusion in Preventing Maternal Hypotension Following Spinal Anesthesia for Caesarean Section
Brief Title: Ephedrine Doses to Prevent Maternal Hypotension After Spinal Anesthesia in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Narottam Jha, Clinical Professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRC/1598/019
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hypotension After Spinal Anesthesia; Hypotension During Cesarean Delivery
MeSH Terms: interventions — Saline Solution; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A who received normal saline immediately after the administration of the (Placebo Comparator): Participants in this group received normal saline immediately after the administration of the subarachnoid block (spinal anesthesia). This group serves as the control group to compare the effectiveness of ephedrine against no pharmacologic intervention
  Interventions: Drug: Normal Saline (Placebo)
- Group B who received ephedrine at a dosage of 1.25 mg/min immediately after the subarachnoid block (Experimental): Participants in this group received ephedrine at a dosage of 1.25 mg/min immediately after the subarachnoid block. This dose is intended to prevent maternal hypotension by maintaining blood pressure during spinal anesthesia.
  Interventions: Drug: Ephedrine
- Group C who received ephedrine at a dosage of 1.5 mg/min immediately after the subarachnoid block (Experimental): Participants in this group received ephedrine at a higher dosage of 1.5 mg/min immediately following the subarachnoid block. This intervention tests whether a slightly higher dose of ephedrine provides better prevention of maternal hypotension without increasing side effects.
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Normal Saline (Placebo) — Participants in the control group receive a continuous intravenous infusion of normal saline, which serves as an inert placebo with no pharmacological effect. This intervention mimics the administration of the active treatments, allowing for direct comparison with the ephedrine groups to assess the effectiveness of the drug in preventing maternal hypotension during spinal anesthesia.
  Arms: Group A who received normal saline immediately after the administration of the
Drug: Ephedrine — The interventions in this study include a control group receiving normal saline, which serves as an inert placebo to assess the effectiveness of the active treatments. Participants in Group B receive an ephedrine infusion at 1.25 mg/min, while those in Group C receive a higher dosage of 1.5 mg/min. This design allows for direct comparison of the two dosages of ephedrine against the control, enabling evaluation of their effectiveness in preventing maternal hypotension following spinal anesthesia during cesarean sections.
  Arms: Group B who received ephedrine at a dosage of 1.25 mg/min immediately after the subarachnoid block
Drug: Ephedrine — The interventions in this study include a control group receiving normal saline, which serves as an inert placebo to assess the effectiveness of the active treatments. Participants in Group B receive an ephedrine infusion at 1.25 mg/min, while those in Group C receive a higher dosage of 1.5 mg/min. This design allows for direct comparison of the two dosages of ephedrine against the control, enabling evaluation of their effectiveness in preventing maternal hypotension following spinal anesthesia during cesarean sections.
  Arms: Group C who received ephedrine at a dosage of 1.5 mg/min immediately after the subarachnoid block

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of different doses of ephedrine infusion in preventing maternal hypotension following spinal anesthesia in parturients undergoing cesarean sections. The study includes 120 participants, aged 18-40 years, with American Society of Anesthesiologists (ASA) physical status II, who are scheduled for elective cesarean delivery. The primary objective is to determine whether low-dose ephedrine infusions at 1.25 mg/min or 1.5 mg/min effectively reduce the incidence of maternal hypotension, with secondary outcomes assessing the need for rescue ephedrine, incidence of side effects (nausea, vomiting, tachycardia), and neonatal Apgar scores. Researchers will compare three groups-saline, 1.25 mg/min ephedrine, and 1.5 mg/min ephedrine-to evaluate their impact on maternal hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cesarean section
* Self-identified as female
* American Society of Anesthesiologists (ASA) physical status II
* Aged between 18 to 40 years
* Full-term singleton pregnancies planned for cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Body mass index (BMI) ≥ 40 kg/m²
* Height less than 145 cm
* Presence of severe neurological or psychiatric conditions
* History of pre-eclampsia
* Severe renal or metabolic disorders
* Contraindications to spinal anesthesia
* Antenatal evidence of fetal anomalies
* Cases with severely compromised fetuses requiring immediate general anesthesia
* Baseline systolic blood pressure (SBP) less than 90 mm Hg
* Pregnancy-induced hypertension
* Refusal to provide written consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is open to individuals who self-identify as female. Eligible participants must be of reproductive age and capable of providing informed consent. The focus on females is due to the study's aim to investigate maternal hypotension during spinal anesthesia specifically in the context of cesarean sections.
Enrollment: 120 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypotension in Patients Undergoing Cesarean Section Following Spinal Anesthesia. | Hypotension episodes were monitored and recorded intraoperatively, immediately following the administration of spinal anesthesia until the end of the cesarean section procedure. The time frame for evaluating this outcome was during the surgical procedure
  The primary outcome of the study is the incidence of maternal hypotension, defined as a decrease in systolic blood pressure (SBP) by more than 20% from baseline, in patients who received different doses of ephedrine (1.25 mg/min or 1.5 mg/min) or saline infusion following spinal anesthesia for cesarean section.

CONTACTS AND LOCATIONS:
Locations (1):
- B.P. koirala Institute of Health Sciences, Dharān, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to researchers upon request. The data will be shared in a de-identified format to protect participant confidentiality.